CLINICAL TRIAL: NCT05310578
Title: Functioning in Individuals with Cervical Radiculopathy After Posterior Cervical Decompression: a Prospective Multicenter Observational Study with a 2 Year Follow-up.
Brief Title: Functioning in Individuals with Cervical Radiculopathy After Posterior Cervical Decompression
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jard Svensson, Physiotherapist, Linkoeping University
Other Study IDs: CR
Record Dates: First submitted 2022-03-03; First posted 2022-04-05 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Posterior cervical foraminotomy (with our without laminectomy) — The aim of surgery is to decrease the compression of the affected nerve. In posterior cervical foraminotomy, the foramina is expanded to create more space and with posterior cervical laminectomy the lamina is removed to create space mainly for the spinal cord.

SUMMARY:
Compression on structures, as spinal nerves, in the cervical spine can cause cervical radiculopathy which leads to pain, disability, and reduced quality of life for the affected individual. Cervical foraminotomy with our without laminectomy are common posterior decompression surgical techniques for treating cervical radiculopathy. There is a lack of knowledge regarding function in patients with cervical radiculopathy after posterior cervical decompression.

The aim with this study is to study pain, function, psychosocial factors, and health related quality of life after posterior cervical decompression in patients with cervical radiculopathy.

This is a prospective multicenter longitudinal observational cohort study with follow-up at three, 12- and 24 months postoperative. A total of 154 individuals scheduled to undergo foraminotomy with our without laminectomy due to cervical radiculopathy will be included. Primary outcome is neck-specific function measured with the Neck Disability Index. Data will be collected preoperatively and at three, 12 and 24 months with electronic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Cervical radiculopathy, confirmed by MRI images (or alternative neuroradiological imaging if MRI contraindicated) compatible with clinical findings of nerve root compression (neurological examination performed by a neurosurgeon/orthopedic surgeon)
* Posterior cervical decompression as foraminotomy with our without laminectomy
* At least 3 months of persistent arm pain
* Age 18-75 years

Exclusion Criteria:

* Nurick score 2 or more (to exclude individuals with moderate to high myelopathy)
* Previous surgery of cervical spine
* Previous fracture or dislocation of the cervical spine
* Malignancy or benign spinal tumor (eg, neuromas)
* Spinal infection
* Previous spondylodiscitis
* Servere mental disorder
* Known alcohol or drug abuse
* Lack of ability to write/comprehend/express oneself in Swedish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cervical radiculopathy scheduled to undergo foraminotomy with our without laminectomy at one of three specific neurosurgery or neuroortopedic clinics in south of Sweden. Individuals are preoperative screened for eligibility and those who meet the criteria to participate in the study are asked for informed consent.
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neck DisabiIity Index; 0-100% (0% = No disability) | Change from baseline to 24 months postoperatively
  To measure neck-specific disability

SECONDARY OUTCOMES:
Numeric Rating Scale; 0-10 (0 = No pain/dizziness) | Change from baseline to 24 months postoperatively
  To measure pain intensity in neck, arm and head; Dizziness and unsteadiness
Frequency of symptoms (5-grade scale from never to always) | Change from baseline to 24 months postoperatively
  To measure frequency of symptoms including neck pain, neck stiffness, headache, arm pain, impaired arm function, dizziness, sleeping problems, visual disturbances, hearing disturbances, difficulty swallowing and chewing, nausea, and problems concentrating.
Specific questions regarding headache and dizziness | Change from baseline to 24 months postoperatively
  To find out more about specific symptoms such as headaches and dizziness
Dizziness Handicap Inventory Scale; 0-100 (0 = no disability) | Change from baseline to 24 months postoperatively
  To measure self-perceived impact on daily life due to dizziness and/or unsteadiness
Short Form Headache Impact test; 36-78 (36 = no impact) | Change from baseline to 24 months postoperatively
  To measure impact of headache in daily life
Core outcome measure Index for neck; 0-10 (0 = good function) | Change from baseline to 24 months postoperatively
  To measure patient self-perceived outcome of spinal surgery
Patient derived Modified Japanese Orthopeadic Association; 0-18 (18 = normal/no myelopathy). | Change from baseline to 24 months postoperatively
  To measure the impact of myelopathy
Odom; 7-point scale (restored/much better to much worse) | Change from baseline to 24 months postoperatively
  To measure global perceived effect
Global rating of change scale; 11 points scale (-5 - 5 where 5 indicates restored). | Change from baseline to 24 months postoperatively
  To measure self-perceived effect
Fear Avoidance Beliefs Questionnaire; 0-96 (0 = no fear). | Change from baseline to 24 months postoperatively
  To measure patients' beliefs about how physical activity and work affect their neck pain
Pain Catastrophizing Scale; 0-52 (0 = no catastrophizing) | Change from baseline to 24 months postoperatively
  To measure catastrophizing
Self-Efficacy Scale; 0-200 (0 = low Self-Efficacy) | Change from baseline to 24 months postoperatively
  To measure confidence in one's own ability
Hospital Anxiety and Depression Scale; 0- 42 (0 = indicates no depression and anxiety) | Change from baseline to 24 months postoperatively
  To measure depression and anxiety
Question regarding expectations of surgery; 4 point scale (restored to no expectation to be restored) | Change from baseline to 24 months postoperatively
  To find out more about expectations of surgery
Cherkin symptom satisfaction | Change from baseline to 24 months postoperatively
  To measure expectations met and satisfaction with care
EuroQuol 5D-5L; 5-25 (5 = high health related quality of life) | Change from baseline to 24 months postoperatively
  To measure health-related quality of life
EQ thermometer; 0-100 (0 = low health related quality of life) | Change from baseline to 24 months postoperatively
  To measure health-related quality of life
Level of physical activity measured with a numeric rating; 1-4 (1 = inactivity - 4 high activity) | Change from baseline to 24 months postoperatively
  To find out more about level of physical activity
International Physical Activity Questionnaire short version (categorize to low, moderate and high activity level) | Change from baseline to 24 months postoperatively
  To measure level of physical activity
Work Ability Index (categorize to poor, moderate, good and excellent work ability) | Change from baseline to 24 months postoperatively
  To measure self-rated work ability

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, PhD, Principal Investigator — Linköping University, Department of Health, Medicine and Caring Sciences, Unit of physiotherapy
Locations (3):
- Sweden (3):
  - Neuro-ortopediska kliniken, Jönköping
  - Neurosurgery clinic, Linköping
  - Ryggkirurgiskt Centrum, Stockholm

IPD SHARING:
Plan to Share IPD: No